CLINICAL TRIAL: NCT05851625
Title: Efficacy of Ear Acupuncture in Preventing Chemotherapy Induced Nausea and Vomiting in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Wahyuningsih Djaali, Lecturer of Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19944
Record Dates: First submitted 2023-04-26; First posted 2023-05-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Cancer; Chemotherapy-induced Nausea and Vomiting; Chemotherapy Effect
Keywords: acupuncture; ear acupuncture; CINV; cancer; press needle
MeSH Terms: conditions — Neoplasms; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The control group was given a placebo press needle acupuncture (using plaster) with standard medical therapy for CINV prevention.
  Interventions: Device: Plesterin
- Acupuncture (Experimental): The intervention group was given press needle acupuncture with standard medical therapy for CINV prevention.
  Interventions: Device: Press needle acupuncture

INTERVENTIONS:
Device: Press needle acupuncture — Press needle acupuncture is a modality of acupuncture using tiny and very thin needles.
  Arms: Acupuncture
Device: Plesterin — The plaster used is a round plaster that resembles the shape of an acupuncture press needle.
  Arms: Placebo

SUMMARY:
Chemotherapy is a cancer therapy performed on advanced cancer with quite good success, but this therapy has quite a lot of side effects. Chemotherapy induced nausea and vomiting or commonly known as CINV, is a condition of nausea and vomiting experienced by cancer patients undergoing chemotherapy, with a prevalence of around 80% of all patients undergoing chemotherapy, and 40% has the potential to become severe. This study aims to determine the efficacy of a new acupuncture modality, namely the press needle, in preventing CINV symptoms in pediatric patients with cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
The study was conducted using a randomized controlled clinical trial (RCT) design in 64 pediatric cancer patients undergoing chemotherapy who were randomized into 2 groups, namely: (1) standard medical therapy as the control group; and (2) a combination of standard therapy with press needle acupuncture as the treatment group. The ear acupuncture points used are Shenmen and Stomach, and one body acupuncture point is PC6. Outcome measurements were carried out in the form of the RINVR questionnaire to assess the intensity of nausea and vomiting measured at 4 times: (1) 12 hours before chemotherapy; (2) 12 hours after chemotherapy; (3) 3 days after chemotherapy; (4) 7 days after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with cancer who are undergoing chemotherapy.
* Age 6 - 18 years.
* Patients with platelet counts > 20,000/μL and neutrophil values > 1,000/μL.
* Willing to follow the research.

Exclusion Criteria:

* Patients with local infection in the puncture area.
* Patients with anatomic abnormalities in the auricle.
* Did not complete the acupuncture therapy until it was finished (three days after chemotherapy).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Rhodes Index of Nausea, Vomiting, and Retching (RINVR) questionnaire | 9 days
  Method instrument for assessing nausea and vomiting consisting of eight statements

CONTACTS AND LOCATIONS:
Overall Officials: Wahyuningsih Djaali, Principal Investigator — Indonesia University
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No